CLINICAL TRIAL: NCT02660047
Title: Magnetic Resonance Assessment of Victoza Efficacy in the Regression of Cardiovascular Dysfunction In Type 2 Diabetes Mellitus and South Asian Descent
Brief Title: Effect of Liraglutide on Cardiovascular Endpoints in Diabetes Mellitus Type 2 Patients of South Asian Descent
Acronym: MAGNA VICTORIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, MalouPaiman, MD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-001623-12
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus Type 2; Metabolic Syndrome; Cardiovascular Disease; Diastolic Dysfunction; Fatty Liver
Keywords: South Asian descent
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Cardiovascular Diseases; Fatty Liver | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Active Comparator): Liraglutide: Solution for subcutaneous injection 6 mg/ml; Flexpen 3 ml.
  Dose: s.c. 0,6 mg (0,1 mL) once daily. After 1 week, the dose will be increased to 1,2 mg (0,2 mL) once daily. If tolerated, after 1 week, dose will be increased to 1.8 mg (0,3 mL) once daily. In case of a hypoglycaemic episode, the dosage of oral blood glucose lowering medicaments will be adjusted first. If hypoglycaemia persists, Liraglutide / Liraglutide placebo will be adjusted on the basis of clinical parameters.
  Duration: 26 weeks
  Interventions: Drug: Liraglutide
- Liraglutide - Placebo (Placebo Comparator): Liraglutide placebo: Solution for injection; Flexpen 3 ml.
  Dose: same as Liraglutide
  Duration: 26 weeks
  Interventions: Drug: Liraglutide - Placebo

INTERVENTIONS:
Drug: Liraglutide — Drug: Liraglutide
  Preparation and labelling of Investigational Medicinal Product:
  Liraglutide will be packed and labeled by Novo Nordisk A/S and provided in non-subject specific boxes. Labeling will be in accordance with Annex 13, local law and trial requirements. The examples of labels are not readily available, but will be supplied when received from Novo Nordisk.
  Drug accountability:
  Drug accountability will be cared for by the Department of Clinical Pharmacy of the LUMC. The trial product will be dispensed to each subject as required according to treatment group by the clinical pharmacist. No trial product will be dispensed to any person not enrolled in the trial.
  Other Names: Trade name: Victoza; EV Product Code: SUB25238; Name of the Marketing Authorisation Holder: Novo Nordisk; Marketing Authorisation number: EU/1/09/529/001; ATC code: A10BX07; CAS number 204656-20-2
  Arms: Liraglutide
Drug: Liraglutide - Placebo — Drug: Liraglutide - Placebo
  Preparation and labelling of Investigational Medicinal Product:
  Liraglutide - Placebo will be packed and labeled by Novo Nordisk A/S and provided in non-subject specific boxes. Labeling will be in accordance with Annex 13, local law and trial requirements. The examples of labels are not readily available, but will be supplied when received from Novo Nordisk.
  Drug accountability:
  Drug accountability will be cared for by the Department of Clinical Pharmacy of the LUMC. The trial product will be dispensed to each subject as required according to treatment group by the clinical pharmacist. No trial product will be dispensed to any person not enrolled in the trial.
  Other Names: Placebo
  Arms: Liraglutide - Placebo

SUMMARY:
Among South Asians, in comparison to Western Europeans, there is an increased risk of type 2 diabetes mellitus (DM2) and DM2-related cardiovascular disease. The effect of Liraglutide (Victoza®) on cardiovascular function is therefore investigated in the DM2 patient group of South Asian descent specifically.

Liraglutide is a new widely prescribed therapeutic agent for DM2 patients. It is a Glucagon Like Peptide - 1 homologue that improves glucose homeostasis and reduces blood pressure and body weight. The disadvantageous metabolic phenotype as seen in South Asians includes a relatively large total fat mass, with predominately visceral relative to subcutaneous adipose tissue and lower brown adipose tissue volume and activity, accompanied by increased lipid levels. The key elements in the mechanism of action of Liraglutide seem to correspond to the differences in metabolic profile between South Asians and Western Europeans. Diastolic dysfunction, an early finding of cardiovascular disease in DM2 and obesity and an independent predictor of mortality, has been shown to be associated with the amount of triglyceride accumulation in the heart and liver. The investigators hypothesize that Liraglutide has direct advantageous cardiovascular effects and reduces triglyceride accumulation in end-organs, specifically for DM2 patients of South Asian descent.

DETAILED DESCRIPTION:
RECRUITMENT AND SCREENING PROCEDURE OF STUDY POPULATION

Patients will be recruited from the outpatient clinics of the Leiden University Medical Center, general practitioners, local hospitals and by advertisement. Patients own physicists will be asked to point eligible patients to the opportunity of study participation. If interested, patients will be informed by the principal investigator. The screening will consist of a medical history, physical examination consisting of measurement of height, body weight, heart rate, blood pressure and examination of thorax and abdomen. Furthermore laboratory tests and rest-ECG will be performed. If the patient is eligible and willing to participate in the study, and has signed the informed consent, the patient will be included. Informed consent must be obtained before any trial related activities take place. After inclusion in the study protocol, the patient's treating physician and general practitioner will be notified.

SAMPLE SIZE CALCULATION

Clinically relevant differences and standard deviations of two studies were chosen to generate data for the sample size calculation. The data we used to incorporate the precision of MRI assessment of cardiac function was generated by a study performed by our group with pioglitazone vs metformin on cardiac function parameters. To estimate the effect of GLP-1 therapy on cardiac function, we only have data of a pilot study with eight DM2 patients with heart failure. With a power of 90% and alfa = 0.05, groups varying from 9 to 17 patients will be needed. In a comparable trial the drop-out rate was 10%. Taken into consideration that the population studied will have a significant better systolic function than the heart failure patients studied by Sokos et al, differences may be smaller. In conclusion, investigators estimate to be able to detect a clinically relevant, significant result with 90% power and alfa = 0.05 with 25 patients in each group.

USE OF CO-INTERVENTION

Patients should continue to use the oral glucose lowering medicaments during the study. For glycaemic control after initiation of the study drug, the current clinical guideline will be followed.

Glycaemic management during study the will be performed as described in appendix 1. To avoid the potential risk of hypoglycaemia, a rigorous monitoring and therapy adjustment schedule will be applied, which will prevent risk of hypoglycemia to a great extent. In addition, patients will be instructed how to recognize and manage a hypo or hyperglycaemic episode. Appropriate individualized adjustments will be made in the unlikely case of a hypo or hyperglycaemic episode. Routine self-measurement of blood glucose by the study participants will be performed once a week. In addition, patients with insulin will be instructed to perform routine self-measurement of blood glucose more frequently when study medication and / or insulin dosage is titrated.

Furthermore patients are asked not to change their diet or level of physical activity during the study period and adequate contraception is obligatory for study participation.

RANDOMIZATION, BLINDING AND TREATMENT ALLOCATION

After the medical screening and mutual agreement of participation in the study, patients will be randomized by block randomization, stratified 1:1 for gender and insulin use. A randomization schedule will be prepared by the research pharmacist who is employee at the Department of Clinical Pharmacy. Coded and sealed envelopes for each participant will be kept at the department of Radiology. In case of safety issues, the sealed envelopes are readily available to the principal investigator and project leader. In case of a serious adverse event - or a medical emergency requiring knowledge of the study medication - the randomization code will be broken. In order to ensure that in medical emergencies, the study participation of the patient is apparent, each patient will receive a patient file in the electronic patient registry. In this personal file, the study number of the patient including the procedure for deblinding and notification of the investigators will be mentioned. When the whole study is completed the randomization list will be provided to the principle investigator by the pharmacist.

STUDY PROCEDURES

Withdrawal of individual subjects: Patients can leave the study at any time for any reason if they wish to do so without any consequences. The responsible investigator can also withdraw a subject if continuing participation is in his opinion deleterious for the subject's wellbeing. Patients can also be withdrawn in case of protocol violations and non-compliance. When a subject withdraws from the study, a medical examination will be performed. In case of withdrawal because of a severe or serious adverse event, appropriate laboratory tests or other special examinations will be performed. Finally patients can be withdrawn from study participation if an incidental finding at the MRI examination - for example a malignancy - influences the ratio of justification versus risks / benefits.

Specific criteria for withdrawal: not applicable

Replacement of individual subjects after withdrawal: Patients will not be replaced after withdrawal, after the first dose of study medication. However, patients may be replaced when withdrawal took place between randomization and administration of the first dose of study medication (for example withdrawal on the first study day due to claustrophobia).

Follow-up of subjects withdrawn from treatment: Follow-up of patients after withdrawal will be done by the treating physicist (general practitioner in most cases). Immediately after study withdrawal, the treating physicist will be updated on the patient's condition and laboratory results and whether the patient was in the control group or intervention group.

Premature termination of the study: In case of the incidence of three serious adverse events, the study will be terminated prematurely and an independent committee will be asked to investigate the safety of the trial. Furthermore, the investigators will prematurely terminate the study when the number of subjects withdrawn from the study exceeds the number used for sample size calculation, i.e. 16 individuals in total.

ADVERSE EVENTS, SERIOUS ADVERSE EVENTS and SUSPECTED UNEXPECTED SERIOUS ADVERSE REACTIONS

Adverse events (AEs):

Adverse events are defined as any undesirable experience occurring to a subject during a clinical trial, whether or not considered related to the used medication or the infused drugs. All adverse events reported spontaneously by the subject or observed by the investigator or his/her staff will be recorded on the adverse event data collection form. The intensity of these adverse events will be graded by the investigator as follows:

* Mild: Discomfort noted but no disruption of normal daily activity
* Moderate: Discomfort sufficient to reduce or affect normal daily activity
* Severe: Inability to work or perform daily activity All adverse events will be actively queried by asking the question: "Have you had any complaints since the last time we talked/met?" at all visits. All adverse events will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated.

The chronicity of the event will be classified by the investigator on a three-item scale as defined below:

* Single occasion: Single event with limited duration
* Intermittent Several episodes of an event, each of limited duration
* Persistent: Event that remains indefinitely

For each adverse event, the relationship to the used medication or infused drug (definite, probable, possible, unknown, definitively not) as judged by the investigator, will be recorded, as well as any actions undertaken in relation to the adverse event, will be recorded. The occurrence of an adverse event that is fatal, life-threatening, disabling or requires in-patient hospitalization, or causes congenital anomaly, will be described according to CHMP guidelines as (suspected) "serious" adverse events and will be notified in writing to the Medical Ethics Committee.

Furthermore, the investigators will copy Novo Nordisk when expediting SARs and SUSARs to competent authorities and will report all SARs related to Novo Nordisk product to Novo Nordisk. The submission to Novo Nordisk must however be within day 15 from the investigator getting knowledge about a valid case no matter local timelines for reporting to the authorities. All pregnancies in trial patients occurring during use of a Novo Nordisk product must be reported to Novo Nordisk.

Serious Adverse Events (SAEs):

A serious adverse event is any untoward medical occurrence or effect that at any dose:

* results in death;
* is life threatening (at the time of the event);
* requires hospitalization or prolongation of existing inpatients' hospitalization;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect;
* Any other important medical event that may not result in death, be life threatening, or require hospitalization, may be considered a serious adverse experience when, based upon appropriate medical judgement, the event may jeopardize the subject or may require an intervention to prevent one of the outcomes listed above.

The sponsor will report the SAEs to the accredited METC that approved the protocol, within 15 days after the sponsor has first knowledge of the serious adverse reactions.

SAEs that result in death or are life threatening should be reported expedited. The expedited reporting will occur not later than 7 days after the responsible investigator has first knowledge of the adverse reaction. This is for a preliminary report with another 8 days for completion of the report.

Suspected Unexpected Serious Adverse Reactions (SUSARs):

Unexpected adverse reactions are SUSARs if the following three conditions are met:

1. the event must be serious
2. there must be a certain degree of probability that the event is a harmful and an - undesirable reaction to the medicinal product under investigation, regardless of the administered dose;
3. the adverse reaction must be unexpected, that is to say, the nature and severity of the adverse reaction are not in agreement with the product information as recorded in:

   * Summary of Product Characteristics (SPC) for an authorized medicinal product;
   * Investigator's Brochure for an unauthorized medicinal product.

The sponsor will report expedited all SUSARs to the competent authorities in other Member States, according to the requirements of the Member States.

The expedited reporting will occur not later than 15 days after the sponsor has first knowledge of the adverse reactions. For fatal or life threatening cases the term will be maximal 7 days for a preliminary report with another 8 days for completion of the report.

SAEs need to be reported till end of study within the Netherlands, as defined in the protocol

STATISTICAL ANALYSIS

Primary and secondary study parameters:

The study endpoints will be analyzed according to intention-to-treat principles. All endpoint parameters are continuous variables. Data will be calculated as mean SD, median (percentile range) according to nature and distribution of the variable. Within group changes from baseline will be tested with independent paired t-test or Wilcoxon signed-rank test. Between group differences will be compared after 26 weeks between Liraglutide and control. Analysis will be performed with SPSS. A 2-sided significance level of p < 0.05 will be applied.

REGULATION STATEMENT

The study will be conducted according to the principles of the "Declaration of Helsinki" (as amended in Tokyo, Venice and Hong Kong, Somerset West and Edinburgh) and in accordance with the Guideline for Good Clinical Practice (CPMP/ICH/135/95 - 17th July 1996).

ADMINISTRATIVE ASPECTS, MONITORING AND PUBLICATION

Handling and storage of data and documents:

Study participants are provided a study name of the letter "MAVI" followed by the number of enrolment (1-50). The study name is coupled to a randomly chosen seven - digit study number. The study number will be used to register the participant in the Electronic Patient Registry of the LUMC. This file will be used as the general patient record, as well as collection of routine laboratory measurements needed for clinical and study treatment. The MRI images will be filed under this registry so that anonymity will be safeguarded. The subject identification code list will be stored by the principal investigator and will only be accessible by the principal investigator and project leader. The data extracted from the study file in the Electronic Patient Registry and from the MRI images will be saved in an SPSS file. From this file the true identity of the study participants can not be discovered. The data will be stored for fifteen years. The blood samples will be frozen and stored anonymously using the above mentioned study name and study number. For ad hoc laboratory tests of inflammatory, endocrine and other biomarkers, blood samples will be kept for a maximum period of three years. The blood samples are solely accessible by the investigator team.

In order to ensure that in medical emergencies, the study participation of the patient is apparent, each patient will receive a patient file in the electronic patient registry. In this personal file, the investigator will mention the study number of the patient including the procedure for de-blinding and notification of the investigators. In this file, the signed Informed Consent form of the patient will be stored.

Public disclosure and publication policy: The data analysis will be performed by the investigators. Novo Nordisk has no role in data analysis and / or publication of the results of the trial in peer reviewed papers. The results of the study will be submitted to peer reviewed papers, also in case the hypothesis has not been proven.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age > 18 years and < 75 years
* BMI > 23 kg/m2
* DM2 treated with metformin and/or SU derivative and/or insulin for at least 3 months in stable dosage
* HbA1c ≥ 6.5% and ≤ 11.0% (≥ 47.5 mmol/mol and ≤ 97.4 mmol/mol)
* EGFR > 30 ml/min
* Ethnicity: South Asian descent (i.e. Hindustani Surinamese), based on self-identified ethnicity and self-reported origin of the mother, the father and the mother's and father's ancestors. Both parents and the mother's and father's ancestors should be South Asian for inclusion.

Exclusion Criteria:

* Use of thiazolidinediones (TZD), GLP-1 analogues, DPP-IV inhibitors, fibrates, prednisone, cytostatic or antiretroviral therapy within 6 months prior to the study
* Uncontrolled treated or untreated hypertension (systolic blood pressue ≥ 180 mmHg and/or diastolic blood pressue ≥ 110 mmHg)
* Acute coronary or cerebrovascular event within 30 days prior to study
* Congestive heart failure NYHA III-IV
* Hereditary lipoprotein disease
* Psychiatric disorders and / or use of antipsychotic or antidepressant drugs at present or in the past
* Hepatic disease (AST/ALT > 2 times reference values)
* Endocrine disease other than diabetes mellitus type 2
* Any significant chronic disease (e.g. inflammatory bowel disease)
* Any significant abnormal laboratory results found during the medical screening procedure
* Gastrointestinal surgery (e.g. gastric bypass)
* Pregnant woman or a woman who is breast-feeding
* Female of child-bearing potential intending to become pregnant or is not using adequate contraceptive methods while sexually active
* Allergy to intravenous contrast
* Known or suspected hypersensitivity to trial products or related products
* Chronic pancreatitis or previous acute pancreatitis
* Personal history or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia type 2
* Claustrophobia
* Metal implants or other contraindications for MRI
* Recent participation in other research projects within the last 3 months or participation in 2 or more projects in one year

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-08; Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Stroke volume | 0 and 26 weeks
  Change from baseline in ml: difference between groups
Ejection Fraction | 0 and 26 weeks
  Change from baseline in percentage: difference between groups
Cardiac output | 0 and 26 weeks
  Change from baseline in L/min: difference between groups
Cardiac index | 0 and 26 weeks
  Change from baseline in L/min/m2: difference between groups
Peak ejection rate | 0 and 26 weeks
  Change from baseline in ml end-diastolic volume/sec: difference between groups
Early peak filling rate | 0 and 26 weeks
  Change from baseline in ml end-diastolic volume/sec: difference between groups
Early deceleration peak | 0 and 26 weeks
  Change from baseline in ml/sec: difference between groups
Atrial peak filling rate | 0 and 26 weeks
  Change from baseline in ml/sec: difference between groups
Early deceleration peak / Atrial peak filling rate (E/A ratio) | 0 and 26 weeks
  Change from baseline of the ratio: difference between groups
Peak mitral annulus longitudinal motion | 0 and 26 weeks
  Change from baseline in cm/sec: difference between groups
Left ventricular filling pressure (= early peak filling rate / peak mitral annulus longitudinal motion) | 0 and 26 weeks
  Change from baseline in mmHg: difference between groups

SECONDARY OUTCOMES:
Aorta vessel wall imaging | 0 and 26 weeks
  Change from baseline of vascular distensibility (pulse wave velocity): difference between groups
Carotid vessel wall imaging | 0 and 26 weeks
  Change from baseline of average vessel wall thickness in mm: difference between groups
Adipose tissue distribution | 0 and 26 weeks
  Change from baseline of the ratio subcutaneous fat / visceral abdominal fat: difference between groups
Total body fat | 0 and 26 weeks
  Change from baseline of total fat volume in ml: difference between groups
Epicardial fat volume | 0 and 26 weeks
  Change from baseline in cm3: difference between groups
Magnetic Resonance Spectroscopy of the heart | 0 and 26 weeks
  Change from baseline in percentage: difference between groups
Magnetic Resonance Spectroscopy of the liver | 0 and 26 weeks
  Change from baseline in percentage: difference between groups
Magnetic Resonance Spectroscopy of the kidney | 0 and 26 weeks
  Change from baseline in percentage: difference between groups
HBA1C | Time Frame: 0,8, 12, 16 and 26 weeks
  Measurements will be used to guide therapeutic management The outcome measure glycemic control will be based on the average HBA1C level of all measurements and regards: difference between groups.
Fasting blood glucose level | 0, 4, 8, 12, 16, 20, 26 weeks
  Fasting blood glucose levels will be used to guide therapeutic management and for safety reasons. Outcome measure: the difference between groups of the average of all measurements.
Myocardial T1 - mapping | 0 and 26 weeks
  Change from baseline of myocardial T1 - values before and after contrast: difference between groups
Brown adipose tissue | 0 and 26 weeks
  Change from baseline of brown adipose tissue volume in cm3: difference between groups

OTHER OUTCOMES:
Anthropometric measurements | 0, 4, 8, 12, 16, 20, 26 weeks
  Length, body weight and calculated BMI. Outcome measure: Change from baseline in kg (body weight) or kg/m2 (BMI): difference between groups
Waist / hip ratio | 0, 4, 8, 12, 16, 20, 26 weeks
  Waist circumference divided by hip circumference. Outcome measure: change from baseline: difference between groups
Systolic blood pressure | 0, 4, 8, 12, 16, 20, 26 weeks
  Measurements for routine clinical management Outcome measure: change from baseline in mmHg: difference between groups
Diastolic blood pressure | 0, 4, 8, 12, 16, 20, 26 weeks
  Measurements for routine clinical management Outcome measure: change from baseline in mmHg: difference between groups
Resting Energy Expenditure | 0, 4, 12, 26 weeks
  Change from baseline: difference between groups Measurement with indirect calorimetry (Jaeger, OxyconPro)
Immunological analysis | 0, 26 weeks
  Fluorescence-Activated Cell Sorting (FACS). Change from baseline: difference between groups.
Immunological analysis | 0, 26 weeks
  Peripheral Blood Mononuclear Cell isolation to analyze immunological activation and status of subjects. Both quantification of white blood cells (T-cells, B-cells, macrophages) and functional analysis will be performed. Change from baseline: difference between groups
Fasting insulin level | 0 and 26 weeks
  Change from baseline: difference between groups
Leptin | 0 and 26 weeks
  Change from baseline: difference between groups
Adiponectin | 0 and 26 weeks
  Change from baseline: difference between groups
CETP | 0, 4, 12 and 26 weeks
  Cholesteryl ester transfer protein Change from baseline: difference between groups
High Sensitive C Reactive Protein | Change from baseline: difference between groups
  0, 4, 12 and 26 weeks
Free Fatty Acids | 0, 4, 12 and 26 weeks
  Change from baseline: difference between groups
Cholesterol level (total, HDL and LDL) | 0, 4, 12 and 26 weeks
  Change from baseline: difference between groups
Liver function tests (ALT, AST, AF, GGT) | 0, 4, 12 and 26 weeks
  Change from baseline: difference between groups
Triglycerides | 0, 4 , 12 and 26 weeks
  Change from baseline: difference between groups
QUICKI | 0 and 26 weeks
  Quantitative Insulin Sensitivity Check Index Change from baseline: difference between groups
Albuminuria | 0 and 26 weeks
  Change from baseline of urinary albumin / creatinine ration: difference between groups
Immunological analysis | 0 and 26 weeks
  Immunological status as assessed by RNA profiling. Change from baseline: difference between groups
Metabolomics | 0 and 26 weeks
  Metabolomics in urine and blood sample. Change from baseline: difference between groups
Insulin dose | 0 and 26 weeks
  Total daily dose (units) of insulin. Change from baseline: difference between groups
Hypoglycaemic episodes | Between week 0 and 26
  Number of grade 1, 2 and 3 hypoglycaemic episodes as detected with self measurement by participants. Comparison between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth HM Paiman, MD, Principal Investigator — Leiden University Medical Center; Huub J van Eyk, MD, Principal Investigator — Leiden University Medical Center; Hildo J Lamb, MD PhD, Study Director — Leiden University Medical Center; Jan W Smit, MD PhD, Study Chair — University Nijmegen Medical Centre; Ingrid M Jazet, MD PhD, Study Chair — Leiden University Medical Center; Albert M de Roos, MD PhD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Albinusdreef 2, Netherlands

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Hoekx CA, Martinez-Tellez B, Straat ME, Bizino MB, van Eyk HJ, Lamb HJ, Smit JWA, Jazet IM, Nahon KJ, Janssen LGM, Rensen PCN, Boon MR. Circulating FGF21 is lower in South Asians compared with Europids with type 2 diabetes mellitus. Endocr Connect. 2025 Jan 6;14(2):e240362. doi: 10.1530/EC-24-0362. Print 2025 Feb 1. PMID 39641307
- [Derived] Straat ME, Martinez-Tellez B, van Eyk HJ, Bizino MB, van Veen S, Vianello E, Stienstra R, Ottenhoff THM, Lamb HJ, Smit JWA, Jazet IM, Rensen PCN, Boon MR. Differences in Inflammatory Pathways Between Dutch South Asians vs Dutch Europids With Type 2 Diabetes. J Clin Endocrinol Metab. 2023 Mar 10;108(4):931-940. doi: 10.1210/clinem/dgac598. PMID 36262060
- [Derived] Dekkers IA, Bizino MB, Paiman EHM, Smit JW, Jazet IM, de Vries APJ, Lamb HJ. The Effect of Glycemic Control on Renal Triglyceride Content Assessed by Proton Spectroscopy in Patients With Type 2 Diabetes Mellitus: A Single-Center Parallel-Group Trial. J Ren Nutr. 2021 Nov;31(6):611-619. doi: 10.1053/j.jrn.2020.09.006. Epub 2020 Dec 5. PMID 33293204
- [Derived] van Eyk HJ, Paiman EHM, Bizino MB, de Heer P, Geelhoed-Duijvestijn PH, Kharagjitsingh AV, Smit JWA, Lamb HJ, Rensen PCN, Jazet IM. A double-blind, placebo-controlled, randomised trial to assess the effect of liraglutide on ectopic fat accumulation in South Asian type 2 diabetes patients. Cardiovasc Diabetol. 2019 Jul 9;18(1):87. doi: 10.1186/s12933-019-0890-5. PMID 31288820